CLINICAL TRIAL: NCT04889222
Title: Effect of Skin Pigmentation and Race/Ethnicity Factors on the Accuracy of Masimo Pulse Oximeters
Status: Terminated | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-21243
Record Dates: First submitted 2021-04-13; First posted 2021-05-17 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- Pulse oximeters (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive pulse oximeter sensors.
  Interventions: Device: INVSENSOR00050; Device: RD SET SpO2

INTERVENTIONS:
Device: INVSENSOR00050 — Noninvasive pulse oximeter sensor
Device: RD SET SpO2 — Noninvasive pulse oximeter sensor

SUMMARY:
This study is designed to compare the accuracy of a noninvasive measurement of oxygen saturation compared to reference values obtained by a laboratory blood gas analyzer. Subgroups will be analyzed by skin pigmentation and self-identified race/ethnicity information.

Study procedures follow ISO-80601-2-61:2011 standard requirements for basic safety and essential performance of pulse oximeter equipment. Arterial blood samples will be collected from subjects while undergoing a controlled desaturation procedure wherein the concentration of oxygen inhaled is slowly reduced until the subject's arterial oxygen concentration is approximately 70%.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 50 years of age.
* Subject weighs a minimum of 110 lbs.
* Subject has a hemoglobin value ≥ 11 g/dL.
* Subject's baseline heart rate is ≥ 45 bpm and ≤ 85 bpm.
* Subject's CO value is ≤ 2.0% FCOHb.
* Subject's blood pressure: Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥ 50 mmHg, and if systolic BP is lower than 100 mmHg and/or diastolic BP is lower than 60 mmHg, subject passes an orthostatic blood pressure test.
* Subject is able to read and communicate in English and understands the study and the risks involved.

Exclusion Criteria:

* Subject is pregnant.
* Subject has a BMI > 35.
* Subject has a history of fainting (vasovagal syncope), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
* Subject has open wounds, inflamed tattoos or piercings, and/or has any visible healing wounds that a medical professional determines may place them at an increased risk for participation.*
* Subject has known drug or alcohol abuse.
* Subject uses recreational drugs.*
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
* Subject has any history of a stroke, myocardial infarction (heart attack), and/or seizures.
* Subject has any chronic bleeding disorder (e.g. hemophilia).
* Subject has taken anticoagulant medication within the past 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
* Subject has donated blood within the past 4 weeks.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject has any symptomatic cardiac dysrhythmia (e.g. atrial fibrillation) and has not received clearance from their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (e.g. schizophrenia, bipolar disorder, multiple sclerosis, Huntington's disease) that interferes with the subject's level of consciousness.*
* Subject has taken opioid pain medication 24 hours before the study.
* Subject has any active signs and/or symptoms of infectious disease (e.g. hepatitis, HIV, tuberculosis, flu, malaria, measles, etc.).*
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year, including but not limited to major dental surgery, appendectomy, plastic surgery, jaw surgery, major ENT surgery, major abdominal and/or pelvic surgery, heart surgery, or thoracic surgery.*
* Subject has symptoms of congestion, head cold, or other illnesses.
* Subject has been in a severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
* Subject has any cancer or history of cancer (not including skin cancer).*
* Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
* Subject is allergic to lidocaine, chlorhexidine, latex, adhesives, or plastic.
* Subject has a heart condition, insulin-dependent diabetes, or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the past 6 months.
* Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis), exercise (working out, riding a bike, riding a skateboard, etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of the investigator/study staff).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulse Oximeters
Started | 54
Completed | 38
Not Completed | 16
Not completed — Did not meet eligibility criteria | 8
Not completed — Failure to place intravenous or arterial line | 3
Not completed — Did not proceed due to time constraints | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pulse Oximeters
Number analyzed (Participants) | 38
Age, Customized [Count of Participants; unit: Participants]
  < 18 years of age | 0
  18 to 50 years of age | 38
  > 50 years of age | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self reported race/ethnicity
  Participants
    Caucasian | 17
    Black or African American | 18
    Hispanic/Black or African American | 1
    Caucasian/Black or African American | 1
    Native American/Black or African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation (SpO2) Accuracy of INVSENSOR00050
Description: Performance of the INVSENSOR00050 sensor will be determined by comparing the noninvasive oxygen saturation measurement (SpO2) of the pulse oximeter sensors to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample and calculating the accuracy root mean square (ARMS) value. The ARMS value will be reported as % of oxygen saturated hemoglobin.
Time Frame: 1-5 hours
Measure: Number; unit: % of oxygen saturated hemoglobin
Arm/Group | Pulse Oximeters
Number analyzed (Participants) | 38
% of oxygen saturated hemoglobin | 1.5

2. Secondary Outcome: Comparison of the Median Bias Between Subgroups for the INVSENSOR00050 Sensor
Description: The secondary outcome is to perform equivalence tests between identified subgroups based on skin pigmentation and/or self-identified race/ethnicity. Since the pulse oximeter displays saturation in integer values, equivalence limits will be set to ± 1% SpO2.
  A TOST procedure using the Wilcoxon Rank Sum Test was used to test the hypothesis that the median biases of the INVSENSOR00050 sensor from two pigmentation subgroups (Light and Dark) were equivalent within ± 1% SpO2. The TOST procedure provides a p-value indicating whether the two measures are equivalent if the p-value is less than 0.05.
Time Frame: 1-5 hours
Population: Due to early termination of the study, the subgroups were not well balanced for secondary outcomes analysis due to lack for female subjects, especially dark skin pigmented females. Hence the analysis is not fully representative. However, the equivalence analysis was conducted for the two pigment subgroups with available data.
Measure: Median (95% Confidence Interval); unit: percentage of SpO2
Arm/Group | Pulse Oximeters
Number analyzed (Participants) | 38
percentage of SpO2
  Dark pigmented subgroup | -0.1 [-0.2 to 0.0]
  Light pigmented subgroup | -1.0 [-1.0 to -0.9]
Statistical Analysis 1: Comparison: Pulse Oximeters; Test type: Equivalence — A TOST procedure using the Wilcoxon Rank Sum Test was used to test the hypothesis that the median biases of the INVSENSOR00050 sensor from two pigmentation subgroups (Light and Dark) were equivalent within ± 1 %SpO2. The TOST procedure provides a p-value indicating whether the two measures are equivalent if the p-value is less than 0.05; p = 0.00097, Two One Sided Tests (TOST) — The a priori threshold for p-value was 0.05

3. Secondary Outcome: Comparison of the Median Bias Between Subgroups for the RD SET SpO2 Sensors
Description: The secondary outcome is to perform equivalence tests between identified subgroups based on skin pigmentation and/or self-identified race/ethnicity. Since the pulse oximeter displays saturation in integer values, equivalence limits will be set to ± 1% SpO2.
  A TOST procedure using the Wilcoxon Rank Sum Test was used to test the hypothesis that the median biases of the RD SET SpO2 sensor from two pigmentation subgroups (Light and Dark) were equivalent within ± 1 %SpO2. The TOST procedure provides a p-value indicating whether the two measures are equivalent if the p-value is less than 0.05.
Time Frame: 1-5 hours
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percentage of SpO2
Arm/Group | Pulse Oximeters
Number analyzed (Participants) | 38
percentage of SpO2
  Dark pigmented subgroup | -0.3 [-0.4 to -0.2]
  Light pigmented subgroup | -0.9 [-1.0 to -0.8]
Statistical Analysis 1: Comparison: Pulse Oximeters; Test type: Equivalence — A TOST procedure using the Wilcoxon Rank Sum Test was used to test the hypothesis that the median biases of the RD SET SpO2 sensor from two pigmentation subgroups (Light and Dark) were equivalent within ± 1 %SpO2. The TOST procedure provides a p-value indicating whether the two measures are equivalent if the p-value is less than 0.05; p = 0.00000, Two One-Sided Tests (TOST) — The a priori threshold for p-value was 0.05

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | Pulse Oximeters
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 1/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pulse Oximeters (N=38)
Blood vessel was potentially damaged during venipuncture. (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT04889222/Prot_SAP_000.pdf